CLINICAL TRIAL: NCT01928537
Title: Phase IIIB, Open-label, Multi-Center Study of the Efficacy and Safety of Rigosertib Administered as 72-hour Continuous Intravenous Infusions in Patients With Myelodysplastic Syndrome With Excess Blasts Progressing On or After Azacitidine or Decitabine
Brief Title: Efficacy and Safety of IV Rigosertib in MDS Patients With Excess Blasts Progressing After Azacitidine or Decitabine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-24; 2013-001124-19 (EudraCT Number)
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2018-07

CONDITIONS: Myelodysplastic Syndromes; Refractory Anemia With Excess Blasts; Chronic Myelomonocytic Leukemia; Cytopenia
Keywords: International Working Group; azacitidine; decitabine
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Cytopenia | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rigosertib sodium (Experimental): Rigosertib sodium will be administered as a 72-hr continuous intravenous infusion consisting of 3 consecutive doses of 1800 mg over 24 hours on Days 1, 2, and 3 of a 14-day cycle for the first 8 cycles and then on Days 1, 2, and 3 of a 28-day cycle for the following cycles.
  Interventions: Drug: rigosertib sodium

INTERVENTIONS:
Drug: rigosertib sodium
  Other Names: ON 01910.Na; SyB L-1101

SUMMARY:
This study will examine the effect intravenously administered rigosertib has on the relationship between bone marrow blasts response and overall survival in myelodysplastic syndromes (MDS) patients who have 5-30% bone marrow blasts and who progressed on or after treatment with azacitidine or decitabine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS confirmed within 6 weeks prior to Screening according to WHO criteria or French-American-British (FAB) classification.
* MDS classified as follows, according to WHO criteria and FAB classification:

  * RAEB-1 (5% to 9% BM blasts)
  * RAEB-2 (10% to 19% BM blasts)
  * CMML (10% to 20% BM blasts) and white blood cells (WBC) < 13,000/μL
  * RAEB-t (20% to 30% BM blasts), meeting the following criteria: WBC < 25,000/μL at study entry; or, Stable White Blood Cell (WBC) at least 4 weeks prior to Screening and not requiring intervention for WBC control with hydroxyurea, chemotherapy, or leukopheresis.
* At least one cytopenia (Absolute Neutrophil Count (ANC) < 1800/μL or Platelet (PLT) count < 100,000/μL or hemoglobin (Hgb) < 10 g/dL).
* Progression (according to 2006 IWG criteria) at any time after initiation of subcutaneous or intravenous azacitidine or decitabine treatment per labeling during the past 2 years, defined as follows:

  * For patients with ˂ 5% BMBL, ≥ 50% increase in BMBL to ˃ 5% BMBL
  * For patients with 5-10% BMBL, ≥ 50% increase in BMBL to ˃ 10% BMBL
  * For patients with 10-20% BMBL, ≥ 50% increase in BMBL to ˃ 20% BMBL
  * For patients with 20-30% BMBL, ≥ 50% increase in BMBL to ˃ 30% BMBL
  * Any of the following: ≥ 50% decrease from maximum remission/response levels in granulocytes or PLT; Decrease in Hgb concentration by ≥ 2 g/dL; or, Transfusion dependence, defined as administration of at least 4 RBC units in the past 8 weeks before Screening (patients must have Hgb values ˂ 9 g/dL prior to transfusion to be considered), in the absence of another explanation.
* Has failed to respond to, relapsed following, not eligible, or opted not to participate in bone marrow transplantation.
* Off all other treatments for MDS for at least 4 weeks, except for azacitidine or decitabine. Filgrastim (G-CSF) and erythropoietin are allowed before and during the study as clinically indicated.
* No medical need for induction chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Patient must signed an informed consent form.

Exclusion Criteria:

* Previous participation in a clinical study of IV or oral rigosertib.
* Anemia due to factors other than MDS (including hemolysis or gastrointestinal [GI] bleeding) unless stabilized for 1 week after RBC transfusion.
* Any active malignancy within the past year, except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast.
* Uncontrolled intercurrent illness including.
* Active infection not adequately responding to appropriate therapy.
* Total bilirubin ≥ 1.5 mg/dL not related to hemolysis or Gilbert's disease.
* ALT/AST ≥ 2.5 x upper limit of normal (ULN).
* Serum creatinine ≥ 2.0 mg/dL.
* Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <130 mEq/L).
* Female patients who are pregnant or lactating.
* Patients who are unwilling to follow strict contraception requirements.
* Female patients with reproductive potential who do not have a negative urine beta-human chorionic gonadotropin (βHCG) pregnancy test at Screening.
* Major surgery without full recovery or major surgery within 3 weeks of Baseline/Cycle 1 Day 1 visit.
* Uncontrolled hypertension (defined as a systolic pressure ≥160 mmHg and/or a diastolic pressure ≥ 110 mmHg).
* New onset seizures (within 3 months prior to Baseline) or poorly controlled seizures.
* Any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy.
* Prior treatment with low-dose cytarabine during the past 2 years.
* Investigational therapy within 4 weeks of Baseline/Day 1 visit.
* Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-08; Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Relationship of bone marrow blast response and overall survival. | Up to 2 years.
  Bone marrow blast response is defined as bone marrow (BM) complete response, ≥ 50% BM blast decrease from pretreatment value, or stable BM response (no progression) according to the International Working Group (IWG) 2006 criteria and overall survival. Overall survival is defined as the time from first study treatment to death from any cause. All patients will be followed until death and/or progression, even if they have discontinued treatment for whatever cause. Survival time of patients lost to follow-up will be censored at the time they were last known to be alive.

SECONDARY OUTCOMES:
Number of patients with overall hematologic response. | Up to 2 years after study enrollment.
  Overall hematologic response (complete remission [CR], partial remission [PR], bone marrow complete response [BMCR], and stable disease [SD]) is defined according to 2006 International Working Group (IWG) response criteria.
Number of patients with hematological improvement. | Up to 2 years after study enrollment.
  Hematological improvement (erythroid response, platelet response and neutrophil response) is defined according to 2006 International Working Group (IWG) response criteria.
Number of patients with cytogenetic response. | Up to 2 years after study enrollment.
  Cytogenetic response is defined according to 2006 International Working Group (IWG) response criteria.
Progression-free survival. | Up to 2 years after study enrollment.
  Progression-free survival is defined as time from date of first dose until date when progression is documented. Progression is defined according to 2006 International Working Group (IWG) response criteria.
Number of patients who transition to Acute Myeloid Leukemia (AML) | Up to 2 years after study enrollment.
  Participants who progress to Acute Myeloid Leukemia (AML) during the study. AML is defined as an increase of at least 50% bone marrow blasts, and more than 20% bone marrow blasts for Refractory Anemia with Excess Blasts types 1 and 2 (RAEB-1 and RAEB-2) and Chronic Myelomonocytic Leukemia (CMML) patients and as an increase of at least 50% bone marrow blasts for Refractory Anemia with Excess Blasts in Transformation (RAEB-t) patients.
Quality of Life Questionnaire | Up to 2 years after study enrollment.
  Change from baseline in responses in the European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire [QLQ]-C30 version 3. Questionnaire will be administered at baseline and at 4 week intervals.
Infections. | Up to 2 years after study enrollment.
  Incidence of infections requiring treatment with intravenous antimicrobials and of bleeding episodes.
Concentration of rigosertib in plasma. | Week 1 and week 3.
  Concentration of rigosertib in plasma will be measured by a validated High Performance Liquid Chromatography (HPLC) method.
Safety. | Study enrollment until 30 days after patient's last dose of rigosertib up to 2 years.
  Counts of patients who have adverse events (AEs). Adverse events will be grouped by system organ class (SOC) and preferred term (PT) using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA), and will be summarized by worst grade according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Fruchtman, MD, Study Chair — Traws Pharma, Inc.
Locations (35):
- United States (14):
  - Stanford University Cancer Center, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Greenbaum Cancer Center University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Texas Southwestern Medical Center-Parkland Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Center, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Denmark (2):
  - Rigshospitalet, Department of Hematology, Copenhagen, Capital Region
  - Aarhus University Hospital, Aarhus, Jylland
- France (2):
  - Hôpital Saint-Louis, Service d'Hématologie, Paris, IDF
  - Institute Paoli Calmettes, Marseille
- Germany (6):
  - Universitätsklinikum Frankfurt, Goethe Universität, Frankfurt am Main, Hesse
  - Universitätsklinikum Köln Klinik I für Innere Medizin, Cologne
  - University Hospital Carl Guslav Carus, Dresden
  - Marien Hospital, Onkologie, Düsseldorf
  - Universitätsmedizin Göttingen, Göttingen
  - Technische Universität München, III. Medizinische Klinik, München
- Italy (3):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - AOU Maggiore della Carità, SCUD Ematologia, Novara
  - Policlinico Umberto 1, Universita "Sapienza", Rome
- Hospital Universitário de Salamanca, Salamanca, Spain
- Sweden (3):
  - Skåne University Hospital,, Lund, Skåne County
  - Sahlgrenska University Hospital, Gothenberg, Västra Götalandsregionen
  - Karolinska University Hospital, Huddinge, Stockholm

REFERENCES:
- [Background] Olnes MJ, Shenoy A, Weinstein B, Pfannes L, Loeliger K, Tucker Z, Tian X, Kwak M, Wilhelm F, Yong AS, Maric I, Maniar M, Scheinberg P, Groopman J, Young NS, Sloand EM. Directed therapy for patients with myelodysplastic syndromes (MDS) by suppression of cyclin D1 with ON 01910.Na. Leuk Res. 2012 Aug;36(8):982-9. doi: 10.1016/j.leukres.2012.04.002. Epub 2012 Apr 21. PMID 22524974
- [Background] Seetharam M, Fan AC, Tran M, Xu L, Renschler JP, Felsher DW, Sridhar K, Wilhelm F, Greenberg PL. Treatment of higher risk myelodysplastic syndrome patients unresponsive to hypomethylating agents with ON 01910.Na. Leuk Res. 2012 Jan;36(1):98-103. doi: 10.1016/j.leukres.2011.08.022. Epub 2011 Sep 14. PMID 21924492
- [Background] Silverman LR, Greenberg P, Raza A, Olnes MJ, Holland JF, Reddy P, Maniar M, Wilhelm F. Clinical activity and safety of the dual pathway inhibitor rigosertib for higher risk myelodysplastic syndromes following DNA methyltransferase inhibitor therapy. Hematol Oncol. 2015 Jun;33(2):57-66. doi: 10.1002/hon.2137. Epub 2014 Apr 29. PMID 24777753
- [Result] Al-Kali A. Relationship of bone marrow blast (BMBL) response to overall survival (OS) in a multicenter study of rigosertib (Rigo) in patients (pts) with myelodysplastic syndrome (MDS) with excess blasts progressing on or after treatment with a hypomethylating agent (HMA). Journal of Clinical Oncology 2017 35:15_suppl, 7056-7056 ASCO 2017
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.